CLINICAL TRIAL: NCT04248049
Title: Clinical Evaluation of Coronal Advanced Flap and Platelet Rich Fibrin on Root Coverage of Gingival Recessions Over a Period of 24 Month.
Brief Title: Platelet Rich Fibrin on Root Coverage of Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Antonio Nariño (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Universidad Antonio Nariño
Record Dates: First submitted 2019-09-04; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Gingival Recession
Keywords: platelet-rich fibrin; platelet concentrates; periodontal diseases
MeSH Terms: conditions — Gingival Recession; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial (RCT) (Interventional)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Split mouth design allowing to evaluate two conditions in the same patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental side (Experimental): Roots covered with coronally advanced flap (CAF) and platelet rich fibrin (PRF) (CAF+PRF)
  Interventions: Other: Platelet rich fibrin
- Control side (Active Comparator): Roots covered with coronally advanced flap (CAR)
  Interventions: Other: Platelet rich fibrin

INTERVENTIONS:
Other: Platelet rich fibrin — The roots of patients with diagnosis of gingival recessions will be covered with coronally advanced flap (CAF) and platelet rich fibrin (PRF) (CAF+PRF)

SUMMARY:
Several surgical techniques and various adjunctive agents have been used to covered Gingival Recession (GR) and promote clinical outcomes. The treatment of the GR more used (gold standard) is the root coverage with surgical procedures and connective tissue graft, but it has limitations due to the conditions of the donor graft. Is necessary develop other biomaterials for these cases.

The platelet rich fibrin is a autologous biomaterial that has gained tremendous momentum having been utilized for a variety of dental and medical procedures including periodontal surgeries. However, results remain contradictory and mainly focus on the hard and soft tissue healing, aesthetics and postoperative discomfort.

The objective of this study was to evaluate the clinical effects of coronal advanced flap (CAF) and CAF + Platelet Rich Fibrin (PRF) on Root coverage (RC) over a period of 24 month.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Healthy males and females of age 18-60 years old
* Multiple bilateral (maxillary or mandibular) gingival recessions (Miller class І or II)
* Good oral hygiene (O´Leary index ≤ 15%)

Exclusion Criteria:

* Active periodontal disease
* Periodontal surgeries in the last three years
* Pregnancy or lactation
* Smokers or alcoholics
* Platelet dysfunction syndrome or thrombocytopenia
* Coagulation defects
* Uncontrolled diabetes
* Medical contraindications to elective oral surgery procedures
* Severe immunodeficiencies
* Oncological history
* Prosthetic restorations adjacent to gingival recessions
* Mobility II or III
* Occlusal contacts excessive
* Root caries
* Buccal restaurations Class V

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change of percentage of root coverage (PRC) from baseline at 12 and 24 months | baseline, 1, 3 , 6, 9, 12 and 24 months
  Complete root coverage after surgical correction measured in percentage by using periodontal probe.
  PRC= Preoperative recession depth - Postoperative recession depth X 100 % Preoperative recession depth

SECONDARY OUTCOMES:
Vertical gingival recession (VGR) | baseline, 1, 3 , 6, 9, 12 and 24 months
  It is measuring the distance from the cemento-enamel junction (CEJ) to the margin of the gingiva at the midbuccal point of the teeth (measured using a periodontal probe in millimeters).
Horizontal gingival recession (HGR) | baseline, 1, 3 , 6, 9, 12 and 24 months
  Measured horizontally between two borders of the recession. (measured using a periodontal probe in millimeters).
Probing depth (PD) | baseline, 1, 3 , 6, 9, 12 and 24 months
  It is measuring the distance from the gingival margin to the base of the pocket using periodontal probe. The probe will be inserted parallel to the long axis of the tooth using light force. (measured using a periodontal probe in millimeters).
Clinical attachment level(CAL) | baseline, 1, 3 , 6, 9, 12 and 24 months
  Two measurements will be used to calculate the CAL: the probing depth and the distance from the gingival margin to the CEJ.
Gingival tissue thickness | baseline, 1, 3 , 6, 9, 12 and 24 months
  The gingiva mid-buccally in the attached gingiva will be penetrated with an endodontic reamer with a silicon disc stop. The measure of penetration will be measured with dentimeter (mm).
Keratinized tissue height (KTH) | baseline, 1, 3 , 6, 9, 12 and 24 months
  To measure the tissue thickness, a guiding device will be made to standardize the region to be measured and then, at a specific point, the mucosa will be punctured with an endodontic spacer and the thickness marked with a rubber marker. Then, using a digital caliper, the thickness will be measured.
Gingival bleeding index (IS) | baseline, 1, 3 , 6, 9, 12 and 24 months
  Evaluation of the presence and absence of bleeding in the gingival margin through the gingival sulcus. The index is calculated after penetration of the sulcus by the periodontal probe, bleeding surfaces are noted and then counted. The index is calculated by dividing the number of surfaces that bleed by the total number of teeth and then multiplying by 100 to reach the percentage of bleeding index.
Visual analog scale (VAS) | baseline, 1, 3 , 6, 9, 12 and 24 months
  Visual analog scale
Evaluation of oral health impact on quality of life, using the Oral Health Impact Profile (OHIP-14) questionnaire. | baseline, 1, 3 , 6, 9, 12 and 24 months
  Evaluate the impact of oral health on patient's quality of life before and 1 year after implant installation. This evaluation will be carried out through the application of a questionnaire with 14 questions (Oral Health Impact Profile: OHIP-14) that assess the patient's perception regarding the impact of oral conditions on their well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Antonio Nariño, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li R, Liu Y, Xu T, Zhao H, Hou J, Wu Y, Zhang D. The Additional Effect of Autologous Platelet Concentrates to Coronally Advanced Flap in the Treatment of Gingival Recessions: A Systematic Review and Meta-Analysis. Biomed Res Int. 2019 Jul 25;2019:2587245. doi: 10.1155/2019/2587245. eCollection 2019. PMID 31428630
- [Background] Debnath K, Chatterjee A. Evaluation of periosteum eversion and coronally advanced flap techniques in the treatment of isolated Miller's Class I/II gingival recession: A comparative clinical study. J Indian Soc Periodontol. 2018 Mar-Apr;22(2):140-149. doi: 10.4103/jisp.jisp_5_18. PMID 29769769
- [Background] Mufti S, Dadawala SM, Patel P, Shah M, Dave DH. Comparative Evaluation of Platelet-Rich Fibrin with Connective Tissue Grafts in the Treatment of Miller's Class I Gingival Recessions. Contemp Clin Dent. 2017 Oct-Dec;8(4):531-537. doi: 10.4103/ccd.ccd_325_17. PMID 29326502
- [Background] Miron RJ, Zucchelli G, Pikos MA, Salama M, Lee S, Guillemette V, Fujioka-Kobayashi M, Bishara M, Zhang Y, Wang HL, Chandad F, Nacopoulos C, Simonpieri A, Aalam AA, Felice P, Sammartino G, Ghanaati S, Hernandez MA, Choukroun J. Use of platelet-rich fibrin in regenerative dentistry: a systematic review. Clin Oral Investig. 2017 Jul;21(6):1913-1927. doi: 10.1007/s00784-017-2133-z. Epub 2017 May 27. PMID 28551729